CLINICAL TRIAL: NCT00459108
Title: A Phase II Trial of Dasatinib (BMS-354825) in Advanced Hepatocellular Carcinoma
Brief Title: Dasatinib in Treating Patients With Advanced Liver Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted early for futility.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00224; NCI-2009-00224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000538220; PHII-83; PHII-83 (Other: City of Hope Medical Center); 7792 (Other: CTEP); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Dasatinib

ARMS (1):
- Oral Dasatinib (Experimental): Patients receive oral dasatinib at 70 mg twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel

SUMMARY:
This phase II trial is studying how well dasatinib works in treating patients with advanced liver cancer that cannot be removed by surgery. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival (PFS) rate and response rate (complete and partial response) at 4 months in patients with unresectable advanced hepatocellular carcinoma treated with dasatinib.

SECONDARY OBJECTIVES:

I. Determine the median PFS and overall survival of patients treated with this drug.

II. Assess the toxicity and tolerability of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3-6 months thereafter.

ELIGIBILITY:
Criteria:

* WBC >= 3,000/mm^3
* LVEF normal
* Histologically or cytologically confirmed hepatocellular carcinoma; Advanced disease, unresectable disease, no Childs C criteria
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* Not a candidate for percutaneous ethanol injection or radiofrequency ablation (RFA)
* Prior transarterial chemoembolization, ethanol, and RFA allowed if new lesions are present in the liver and there are no other sites of disease
* No pleural effusion or ascites requiring paracentesis within the past 4 weeks
* No known brain metastases
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 3 months
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 75,000/mm^3
* Bilirubin =< 2 times upper limit of normal (ULN)
* AST and ALT =<2.5 times ULN (5 times ULN if liver involvement by tumor)
* Creatinine =< 2 times ULN
* PT =< 1.5 times ULN (no anticoagulation)
* Albumin >= 2.5 mg/dL
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to dasatinib
* No evidence of encephalopathy
* No condition that would preclude ability to swallow and retain dasatinib tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication;
  * Requirement for IV alimentation;
  * Prior surgical procedures affecting absorption:
  * Active peptic ulcer disease
* No clinically significant ECG abnormalities
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction or ventricular tachyarrhythmia within the past 6 months;
  * Prolonged QTc >= 480 msec (Fridericia correction);
  * Major conduction abnormality (unless cardiac pacemaker is present)
* No other uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection;
  * History of significant bleeding disorder, including congenital (von Willebrand's disease) or acquired disorders (antifactor VIII antibodies);
  * Psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from all prior therapy
* One prior systemic chemotherapy regimen allowed
* Prior cryosurgery allowed
* More than 4 weeks since prior transarterial chemoembolization
* More than 4 weeks since prior radiotherapy
* Prior or concurrent localized palliative radiotherapy (i.e., bony metastasis) allowed provided it was administered for =< 3 days
* At least 7 days since prior and no concurrent antithrombotic and/or antiplatelet agents (e.g., warfarin, heparin, low molecular weight heparin, acetylsalicylic acid, and/or ibuprofen)
* At least 7 days since prior and no concurrent agents with proarrhythmic potential
* At least 7 days since prior and no concurrent medications or substances that are potent inhibitors or inducers of CYP3A4
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent embolization or chemoembolization
* No concurrent systemic antacids (H2 receptor antagonists or proton pump inhibitors)
* Locally active antacids allowed provided they are held for 2 hours before and 2 hours after dasatinib dose
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — City of Hope Medical Center
Locations (1):
- University of Southern California, Norris, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Dasatinib: Patients receive oral dasatinib twice daily at 70 mg on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  dasatinib: Given orally
Period: Overall Study
Arm/Group | Oral Dasatinib
Started | 25
Completed | 14
Not Completed | 11
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 61 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Response = CR + PR
Time Frame: 4 months
Measure: Number; unit: percentage of responding patients
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
percentage of responding patients | 0

2. Primary Outcome: Four Month Progression-free Survival (PFS)
Description: Progression-free survival calculated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
percentage of participants | 40 [21 to 58]

3. Secondary Outcome: Median Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression or death, up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
Months | 3.7 [1.8 to 6.4]

4. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
Months | 7.5 [2.9 to 13.6]

5. Secondary Outcome: Safety and Tolerability
Description: Summarize observed grade 3 and higher toxicities related to dasatanib. The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 were used for reporting.
Time Frame: Up to 4 years
Population: One patient died due to underlying cardiac disease which may have been exacerbated by the dasatanib.
Measure: Number; unit: participants
Arm/Group | Oral Dasatinib
Number analyzed (Participants) | 25
participants
  Grade 3 : AST, SGOT | 2
  Grade 3 : Anorexia | 2
  Grade 3 : Sudden death | 0
  Grade 3 : Dehydration | 2
  Grade 3 : Diarrhea | 1
  Grade 3 : Dizziness | 0
  Grade 3 : Edema:head and neck | 1
  Grade 3 : Fatigue (asthenia, lethargy, malaise) | 8
  Grade 3 : Glucose, serum-high (hyperglycemia) | 1
  Grade 3 : Hemoglobin | 2
  Grade 3 : Hemorrhage, GI - Colon | 1
  Grade 3 : Hemorrhage, GI - Stomach | 1
  Grade 3 : Infection with normal ANC | 1
  Grade 3 : Leukocytes (total WBC) | 1
  Grade 3 : Lymphopenia | 2
  Grade 3 : Nausea | 3
  Grade 3 : Pain - Head/headache | 2
  Grade 3 : Pain - Middle ear | 1
  Grade 3 : Phosphate, serum-low (hypophosphatemia) | 3
  Grade 3 : Platelets | 1
  Grade 3 : Pneumonitis/pulmonary infiltrates | 1
  Grade 3 : Potassium, serum-low (hypokalemia) | 1
  Grade 3 : Proteinuria | 1
  Grade 3 : Sodium, serum-low (hyponatremia) | 3
  Grade 3 : Thrombotic microangiopathy | 1
  Grade 3 : Urinary retention | 1
  Grade 3 : Vomiting | 3
  Grade 4 : AST, SGOT | 0
  Grade 4 : Anorexia | 0
  Grade 4 : Sudden death | 0
  Grade 4 : Dehydration | 0
  Grade 4 : Diarrhea | 0
  Grade 4 : Dizziness | 1
  Grade 4 : Edema:head and neck | 0
  Grade 4 : Fatigue (asthenia, lethargy, malaise) | 1
  Grade 4 : Glucose, serum-high (hyperglycemia) | 0
  Grade 4 : Hemoglobin | 1
  Grade 4 : Hemorrhage, GI - Colon | 0
  Grade 4 : Hemorrhage, GI - Stomach | 0
  Grade 4 : Infection with normal ANC | 0
  Grade 4 : Leukocytes (total WBC) | 0
  Grade 4 : Lymphopenia | 0
  Grade 4 : Nausea | 0
  Grade 4 : Pain - Head/headache | 0
  Grade 4 : Pain - Middle ear | 0
  Grade 4 : Phosphate, serum-low (hypophosphatemia) | 0
  Grade 4 : Platelets | 0
  Grade 4 : Pneumonitis/pulmonary infiltrates | 0
  Grade 4 : Potassium, serum-low (hypokalemia) | 0
  Grade 4 : Proteinuria | 0
  Grade 4 : Sodium, serum-low (hyponatremia) | 0
  Grade 4 : Thrombotic microangiopathy | 0
  Grade 4 : Urinary retention | 0
  Grade 4 : Vomiting | 0
  Grade 5 : AST, SGOT | 0
  Grade 5 : Anorexia | 0
  Grade 5 : Sudden death | 1
  Grade 5 : Dehydration | 0
  Grade 5 : Diarrhea | 0
  Grade 5 : Dizziness | 0
  Grade 5 : Edema:head and neck | 0
  Grade 5 : Fatigue (asthenia, lethargy, malaise) | 0
  Grade 5 : Glucose, serum-high (hyperglycemia) | 0
  Grade 5 : Hemoglobin | 0
  Grade 5 : Hemorrhage, GI - Colon | 0
  Grade 5 : Hemorrhage, GI - Stomach | 0
  Grade 5 : Infection with normal ANC | 0
  Grade 5 : Leukocytes (total WBC) | 0
  Grade 5 : Lymphopenia | 0
  Grade 5 : Nausea | 0
  Grade 5 : Pain - Head/headache | 0
  Grade 5 : Pain - Middle ear | 0
  Grade 5 : Phosphate, serum-low (hypophosphatemia) | 0
  Grade 5 : Platelets | 0
  Grade 5 : Pneumonitis/pulmonary infiltrates | 0
  Grade 5 : Potassium, serum-low (hypokalemia) | 0
  Grade 5 : Proteinuria | 0
  Grade 5 : Sodium, serum-low (hyponatremia) | 0
  Grade 5 : Thrombotic microangiopathy | 0
  Grade 5 : Urinary retention | 0
  Grade 5 : Vomiting | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 3 years, 3 months.
Description: "Other" adverse events include all grades and attributions to treatment not included in the "Serious" adverse event table.
Arm/Group | Oral Dasatinib
Serious Adverse Events (participants affected / at risk) | 13/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Dasatinib (N=25)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 3 (3)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Prostatic hemorrhage (Reproductive system and breast disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Dasatinib (N=25)
Hemoglobin decreased (Blood and lymphatic system disorders) | 16 (43)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Dry eye syndrome (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 11 (18)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 10 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 13 (26)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (16)
Chest pain (General disorders) | 1 (2)
Chills (General disorders) | 3 (4)
Disease progression (General disorders) | 16 (16)
Edema limbs (General disorders) | 8 (10)
Fatigue (General disorders) | 15 (41)
Fever (General disorders) | 8 (12)
Localized edema (General disorders) | 3 (4)
Pain (General disorders) | 6 (9)
Hepatic pain (Hepatobiliary disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 1 (3)
Infection (Infections and infestations) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 14 (35)
Alkaline phosphatase increased (Investigations) | 13 (25)
Aspartate aminotransferase increased (Investigations) | 15 (40)
Bilirubin increased (Investigations) | 6 (11)
Creatinine increased (Investigations) | 7 (13)
Leukocyte count decreased (Investigations) | 7 (18)
Lipase increased (Investigations) | 2 (12)
Lymphocyte count decreased (Investigations) | 6 (10)
Neutrophil count decreased (Investigations) | 5 (15)
Platelet count decreased (Investigations) | 10 (26)
Weight loss (Investigations) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 12 (23)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 6 (15)
Blood glucose increased (Metabolism and nutrition disorders) | 9 (27)
Dehydration (Metabolism and nutrition disorders) | 5 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 9 (12)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 8 (14)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 12 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 13 (21)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Sinus pain (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 4 (6)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 4 (13)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (14)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less